CLINICAL TRIAL: NCT00103519
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled Study of DITPA in Patients With NYHA Class III and IV Congestive Heart Failure Who Have Low Serum T3 Levels
Brief Title: Study of DITPA in Patients With Congestive Heart Failure
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated for reasons unrelated to safety or efficacy.
Sponsor: Titan Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DIT-803
Record Dates: First submitted 2005-02-09; First posted 2005-02-10 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2006-11

CONDITIONS: Heart Failure, Congestive
Keywords: Heart Failure, DITPA
MeSH Terms: conditions — Heart Failure | interventions — 3,5-diiodothyropropionic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- DITPA 180 mg/day (Experimental): DITPA 180 mg/day BID
  Interventions: Drug: DITPA (3,5-diiodothyropropionic acid)
- DITPA 360 mg/day (Experimental): DITPA 360 mg/day BID
  Interventions: Drug: DITPA (3,5-diiodothyropropionic acid)
- Placebo (Placebo Comparator): Placebo BID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DITPA (3,5-diiodothyropropionic acid)
  Arms: DITPA 180 mg/day; DITPA 360 mg/day
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study will assess the safety and efficacy of DITPA relative to placebo in patients with New York Heart Association (NYHA) class III or IV congestive heart failure (CHF) who have low serum T3. DITPA is an investigational agent.

DETAILED DESCRIPTION:
Rationale: Congestive heart failure (CHF) is a major public health problem associated with significant morbidity and mortality in patients with New York Heart Association (NYHA) class III or IV disease. Multiple studies have identified a particularly high-risk group of patients who have reduced thyroid hormone activity, specifically, low serum triiodothyronine (T3) levels. This group represents approximately 30% of patients with NYHA class III or IV disease and has significantly higher mortality rates than those with normal T3.

DITPA (3,5-diiodothyropropionic acid) is an analogue of naturally occurring thyroid hormone (T3) that has been specifically designed to improve cardiac performance with a lower potential for tachycardia in CHF patients. Although structurally similar to T3, DITPA has a propionic acid side chain and lacks an iodine at the 3' position of the outer phenolic ring. While DITPA binds to the same thyroid hormone receptors as T3, binding affinities are significantly less, suggesting partial agonistic actions. Preclinical studies with DITPA have supported a rationale for its use in patients with CHF.

Primary objective: To assess the safety and tolerability of DITPA in patients with NYHA class III/IV CHF and low serum T3.

Secondary Objective: To obtain preliminary evidence of the efficacy of DITPA in patients with NYHA class III/IV CHF and low serum T3

Design: The multi-center, randomized, double-blind, placebo-controlled study is designed to evaluate the safety and tolerability of DITPA in patients with NYHA class III or IV CHF who have low levels of serum T3 with normal levels of thyroid stimulating hormone (TSH).

One hundred and fifty patients at approximately 35 centers in the U.S. will be randomized to 1 of 3 treatment groups in a 1:1:1 ratio (i.e., 50 patients per treatment group):

* DITPA at 180 mg/day (90 mg twice a day [BID], orally)
* DITPA at 360 mg/day (180 mg BID, orally)
* Placebo BID, orally

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 18 years of age
* NYHA class III or IV CHF
* Females must not be pregnant or lactating. Females of childbearing potential and males must use a reliable means of contraception
* Serum total T3 <= 95 ng/dL with normal levels of TSH
* On a regimen consisting of angiotensin-converting enzyme inhibitors and/or angiotensin receptor antagonists, beta blockers, and diuretics for a minimum of 3 months prior to randomization
* Clinically stable for 2 weeks prior to randomization (defined as no change in functional class by NYHA, no hospitalization or ER visit, and no intravenous inotropic or vasodilator treatment for 2 weeks)
* An LVEF <= 40%, documented within 6 months prior to randomization, or > 6 months with confirmation of LVEF by local echocardiographic measurements within 2 weeks prior to randomization
* Able to give informed consent

Exclusion Criteria:

* New onset CHF (less than 3 months prior to randomization)
* Active myocarditis, hypertrophic cardiomyopathy, uncorrected primary valvular disease, restrictive cardiomyopathy, uncorrected congenital heart disease, or constrictive pericarditis
* Myocardial infarction, unstable ischemic heart disease, stroke, or coronary revascularization procedure within 4 weeks prior to randomization; or an expectation of a coronary revascularization procedure, cardiac transplant, or left ventricular assist device placement being needed within 24 weeks after randomization
* History of sudden arrhythmic syncope or sustained ventricular arrhythmia, unless the patient has an implantable cardioverter defibrillator (ICD) for at least 12 weeks prior to randomization; history of clinically significant heart block, unless the patient has had a pacemaker at least 12 weeks prior to randomization
* History of cardiac resynchronization therapy in the last 12 weeks prior to randomization or expectation of cardiac resynchronization therapy or ventricular mechanical assistance needed within 24 weeks after randomization
* History of cardiac transplant
* Heart rate < 50 beats per minute or > 130 beats per minute
* Systolic blood pressure <= 80 mm Hg
* Serum creatinine => 2.5 mg/dL
* Treatment with intravenous vasodilators (including nesiritide) or inotropes within 2 weeks prior to randomization
* Receipt of any other investigational agent or device within 4 weeks prior to randomization
* Diagnosis of other non-cardiac underlying medical conditions expected to impact their mortality within 24 weeks after randomization
* Drug or alcohol dependence, or other conditions which may affect study compliance
* History of thyroid disorders of any form within 24 weeks prior to randomization
* Use of thyroid supplements (levothyroxine, liothyronine, etc.) or any preparation containing thyromimetic agents within 24 weeks prior to randomization
* Supraventricular arrhythmia refractory to conventional treatment, as judged by the investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2004-12; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of DITPA

SECONDARY OUTCOMES:
Efficacy of DITPA

CONTACTS AND LOCATIONS:
Overall Officials: Milton Packer, MD, Study Chair — University of Texas Southwestern Medical Center
Locations (22):
- United States (22):
  - The Heart Center, Huntsville, Alabama
  - Cardiac Solutions, Peoria, Arizona
  - University of Arizona Sarver Heart Center, Tucson, Arizona
  - University of Southern California, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Cardiovascular Consultants Medical Group, Walnut Creek, California
  - Saint Joseph's Research Institute, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Louisville, Louisville, Kentucky
  - Louisiana State University Health Science Center, Shreveport, Louisiana
  - Mayo Clinic, Rochester, Minnesota
  - Columbia University New York Presbyterian Hospital, New York, New York
  - Cincinnati VA Medical Center, Cincinnati, Ohio
  - Clevaland Clinic Foundation, Cleveland, Ohio
  - Oklahoma Foundation for Cardiovascular Research, Oklahoma City, Oklahoma
  - Oregon Health Sciences University, Portland, Oregon
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Baylor University Medical Center Heart Place, Dallas, Texas
  - The University of Virginia Health System, Charlottesville, Virginia
  - William S. Middleton Memorial Veterans Hospital, Madison, Wisconsin